CLINICAL TRIAL: NCT01000519
Title: Differential Effects of Aerobic Versus Progressive Resistance Training on Metabolic Profile and Fitness in Older Adults With Diabetes Mellitus - a Randomized Controlled Trial
Brief Title: Effects of Different Mode of Exercise Training on Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRC/0728/2003
Record Dates: First submitted 2009-10-20; First posted 2009-10-23 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus; Randomized control trial; Exercise; Hemoglobin A, Glycosylated
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity | interventions — Exercise Test; Resistance Training; Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Training (Active Comparator): 50 minutes of aerobic training, 18 sessions within 2 months period
  Interventions: Other: Aerobic Training
- Progressive Resistance Training (Experimental): 50 minutes of progressive resistance training consisting of nine resistance exercises, each conducted 3 sets of 10 repetitions. 18 sessions over 2 months period.
  Interventions: Other: Progressive resistance training

INTERVENTIONS:
Other: Aerobic Training — 18 sessions over 2 months period. Each session consist of 50 minutes of aerobic training at 65-70 % of maximum predicted heart rate
  Other Names: Treadmill; Cross trainer; Cycling
  Arms: Aerobic Training
Other: Progressive resistance training — 18 sessions completed in 2 months. each session consists of 50 minutes of resistance training which is made up of 3 sets of 10 repetitions of nine resistive exercises using machines and free weights at 65-70% of 1-repetitive maximum.
  Other Names: Weight training; Circuit training
  Arms: Progressive Resistance Training

SUMMARY:
Randomized study on the comparison between aerobic training versus progressive resistance training over a 2 months period for older adults with type 2 diabetes. The hypothesis is that progressive resistance training is just as effective as aerobic training on Hba1c and could be an alternative training for those older diabetic patients who cannot participate in aerobic exercise.

DETAILED DESCRIPTION:
Many studies have shown the importance of aerobic training with respect to management of diabetes. However adoption of aerobic activities may be challenging for some individuals with diabetes, especially the elderly and the obese. There is increasing interest in resistance training and no study have looked at direct comparison between the two.

Subjects with diabetes but is generally sedentary (determined by means of a questionnaire) were recruited and randomized in one of the two groups. Subjects are supervised in a group and a completer is defined as one who completed 18 sessions within 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 years and above,
* Hba1c between 8 to 10 % in the past one month,
* sedentary,
* able to continuously walk for at least 20 minutes and climbed one flight of stairs unaided without stopping were eligible for participation.

Exclusion Criteria:

* uncontrolled diabetes mellitus with Hba1c more than 10% or if escalation of treatment of glycemic control or dyslipidemia was likely to be necessary over the 2 months training period period,
* congestive cardiac failure, unstable angina or acute myocardial infarction within the last one year,
* proliferative diabetic retinopathy,
* uncontrolled hypertension,
* advanced arthritis likely to limit mobility or participation in prescribed exercises,
* respiratory conditions such as asthma and chronic obstructive lung disease,
* significant proteinuria or chronic renal insufficiency,
* received drugs for the treatment of obesity or very low caloric diet (VLCD, less than 1000 kcal/ day),
* renal disease and
* inability to monitor glucose level or comply with exercise program.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-12; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A, Glycosylated (Hba1c). Measuring unit: percentage | 2 months
  Blood was drawn from each subject who fasted at least 10 hours overnight. Hba1c (%) was measured using high performance liquid chromatography (HPLC Variant II Bio Rad Laboratories, Munich, Germany). Change in Hba1c before and after intervention were looked at.

SECONDARY OUTCOMES:
Peak volume of oxygen consumed (VO2peak) or fitness level. Measuring unit: ml/kg/min | 2 months
  Modified Bruce protocol on a treadmill using Cosmed K4B2 machine to measure
Anthropometric measurements | 2 months
  weight (kilogram), height (metres), body mass index (BMI), waist circumference (centimeters) and body fat (percentage). Measurements to be taken before and after intervention.
Cholesterol | 2 months
  Blood was drawn from each subject who fasted at least 10 hours overnight. Total cholesterol and triglycerides (TG) were measured using enzymatic colorimetric methods with cholesterol oxidase-peroxidase amino phenazone phenol and glycerol-3-phospahte oxidase-peroxidase amino phenazone phenol. High-density lipoprotein cholesterol (HDL-C) was measured using homogenous enzymatic colorimetric assay. Low-density lipoprotein cholesterol (LDL-C) was calculated using the Friedewald formula.

CONTACTS AND LOCATIONS:
Overall Officials: Li Whye Cindy Ng, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Background] Arora E, Shenoy S, Sandhu JS. Effects of resistance training on metabolic profile of adults with type 2 diabetes. Indian J Med Res. 2009 May;129(5):515-9. PMID 19675378
- [Derived] Ng CL, Tai ES, Goh SY, Wee HL. Health status of older adults with Type 2 diabetes mellitus after aerobic or resistance training: a randomised trial. Health Qual Life Outcomes. 2011 Aug 2;9:59. doi: 10.1186/1477-7525-9-59. PMID 21810269
- [Derived] Ng CL, Goh SY, Malhotra R, Ostbye T, Tai ES. Minimal difference between aerobic and progressive resistance exercise on metabolic profile and fitness in older adults with diabetes mellitus: a randomised trial. J Physiother. 2010;56(3):163-70. doi: 10.1016/s1836-9553(10)70021-7. PMID 20795922